CLINICAL TRIAL: NCT04572555
Title: The Effects of Heat Application on Depression, Anxiety, Menstrual Attitude and Severity of Dysmenorrhea at 4 Menstrual Cycle
Brief Title: Heat Application on Depression, Anxiety, Menstrual Attitude and Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Hülya TÜRKMEN, Lecturer (PhD), Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BalıkesirM
Record Dates: First submitted 2020-09-23; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: DYSMENORRHEA
Keywords: Dysmenorrhea; Heat Treatment; Depression Anxiety, Stress; Menstrual Attitude
MeSH Terms: conditions — Dysmenorrhea; Fever | interventions — Diathermy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat Treatment Group (Experimental): Thermoforming was applied to the lower abdomen by the subjects themselves when the dysmenorrhea pain was at its peak. The subjects were instructed on the application of the thermophores. Thermoforming was applied wrapped in towels in order to shield the subjects from the effects of direct heat. In a study, heat packs that had a temperature of 38.9 °C were used for treatment of dysmenorrhea. In this study, the temperature of the water used in the thermoforming process was 45 °C. Considering the risk of the thermophores cooling down and the shielding provided by the towels, the water temperature was kept higher compared to those in other studies. The temperature of the water was measured using a liquid thermometer. Heat treatment was applied for 20 minutes without interruptions.
  Interventions: Other: Heat Treatment
- Control Group (No Intervention): No Intervention

INTERVENTIONS:
Other: Heat Treatment — Thermoforming was applied to the lower abdomen by the subjects themselves when the dysmenorrhea pain was at its peak.
  Arms: Heat Treatment Group

SUMMARY:
AIM: Establishing the effects of heat application on depression, anxiety, menstrual attitude and severity of dysmenorrhea.

METHODS: This randomized controlled prospective experimental trial was conducted with 43 students who were suffering from dysmenorrhea under 2 groups, the heat treatment group (n=20) and the control group (n=23). To the heat treatment group, dry heat was applied for 20 minutes to the lower abdominal region of the subjects when their dysmenorrhea was most severe. The control group did not receive any treatments. The data were acquired by using a Personal Information Form. The Visual Analogue Scale (VAS) for determining the severity of dysmenorrhea, the Short Form McGill Pain Questionnaire to establish the type of pain, the Menstrual Attitude Questionnaire to establish the attitude and the practices during dysmenorrhea and the Depression Anxiety and Stress Scale to determine the psychological impacts of dysmenorrhea were used. In the first menstrual cycle, both groups received the questionnaires, and no treatment was applied. At the second, third and fourth menstrual cycles, VAS and the McGill Pain Questionnaire were applied before the treatment (T1), right after the treatment (T2) and 2 hours after the treatment (T3). The Menstrual Attitude Questionnaire and the Depression Anxiety and Stress Scale were applied right after the treatment.

DETAILED DESCRIPTION:
This experimental randomized controlled prospective study was conducted at the tocology department of a university hospital in Balikesir, Turkey between March 2019 and June 2019.

The sample size was determined using G * Power 3 calculations in accordance with prior studies on heat application to the lower abdomen. Estimation of the effects was acquired from the findings of Potur and Kömürcü (2014), who reported a pain severity of 1.99 ± 2.42 in the heat-treated group and 5.78 ± 2.63 in the control group. We aimed to establish a similar difference. For each group, the sample count was determined as 12. However, in order to increase the power of the study, 23 students were included both in the heat treatment group and the control group, totaling up to 46 individuals for the sample. Power analysis indicated that the size of the sample had a power of 96% with α = 0.05. The decrease comparative to the control group in the severity of dysmenorrhea pain after heat application had an effect size of 0.616.

The inclusion criteria were determined as being at the ages of 18-30, being nulliparous, having a VAS score of 2 and higher [24], not having a systemic or chronic disease and not using hormonal contraceptives. The exclusion criteria were determined as using forms of analgesic and alternative treatments during the study (1 subject in the heat treatment group was excluded at the 3rd menstrual cycle) and experiencing menstrual irregularities (3 subjects in the heat treatment group and 4 subjects in the control group were excluded at the 3rd menstrual cycle).

To the sample of the study, students with dysmenorrhea pain were admitted. Randomization was achieved by having the subjects pull envelopes for the designation of their groups. Students who pulled the 'Heat Treatment Group' were allocated to the heat treatment group, and the students who pulled the 'Control Group' were allocated to the control group. A total of 46 students partook in the study, and 3 students from the heat treatment group were excluded from the study by their own requests. At the 1st and the 2nd menstrual cycles, the heat treatment group consisted of 20 subjects, and the control group consisted of 23. At the 3rd menstrual cycle, 4 subjects from the heat treatment group and 4 subjects from the control group were excluded from the study in accounts of their analgesic medicine usage or inability to menstruate. At the 3rd and 4th menstrual cycles, the heat treatment group had 16 subjects, and the control group had 19.

For the collection of the data, Personal Information Forms were developed by the researchers in accordance with the scientific literature, the Visual Analogue Scale (VAS) in order to establish the severity of the dysmenorrhea pain, the Short Form McGill Pain Questionnaire to determine the types of pain, the Menstrual Attitude Questionnaire to establish the attitudes and the behaviors during menstruation and the Depression Anxiety and Stress Scale to determine the psychological effects of dysmenorrhea were utilized. The Personal Information Form was applied to the heat treatment group and the control group after receiving permission from the subjects. The subjects were observed for a total of 4 menstrual cycles. The subjects in the heat treatment group and the control group were instructed not to use any analgesic medication or alternative treatments during the study. In the 1st menstrual cycle, heat treatment was not applied to the subjects. In the first menstrual cycle, the Short Form McGill Pain Questionnaire, VAS, the Menstrual Attitude Questionnaire and the Depression Anxiety and Stress Scale was applied at the peak severity of dysmenorrhea pain. In the following 3 menstruation cycles, VAS-T1 and the Short Form McGill Pain Questionnaire-T1 were applied to the heat treatment group and the control group at the peak severity of dysmenorrhea pain. Later, 20 minutes of heat treatment was applied to the heat treatment group. The control group were not given any treatments. VAS-T2, the Short Form McGill Pain Questionnaire-T2, the Menstrual Attitude Questionnaire and the Depression Anxiety and Stress scale were applied to the subjects in both groups 20 minutes after the primary evaluation. VAS-T3 and the Short Form McGill Pain Questionnaire were applied to both groups 2 hours after the primary evaluation.

Thermoforming was applied to the lower abdomen by the subjects themselves when the dysmenorrhea pain was at its peak. The subjects were instructed on the application of the thermophores. Thermoforming was applied wrapped in towels in order to shield the subjects from the effects of direct heat. In a study, heat packs that had a temperature of 38.9 °C were used for treatment of dysmenorrhea. In this study, the temperature of the water used in the thermoforming process was 45 °C. Considering the risk of the thermophores cooling down and the shielding provided by the towels, the water temperature was kept higher compared to those in other studies. The temperature of the water was measured using a liquid thermometer. Heat treatment was applied for 20 minutes without interruptions.

Visual Analogue Scale (VAS): This scale was utilized to establish the severity of the dysmenorrhea pain in the subjects. The scale consists of a 10 cm vertical line starting with 0 and ending with 10. In this study, VAS was applied in 4 menstrual cycles; 1st menstrual cycle, once when the pain was most severe (T1), at the 2nd, 3rd and the 4th menstrual cycles, once when the pain was most severe (T1), 20 minutes after the primary application (T2) and 2 hours after the first application (T3).

Short Form McGill Pain Questionnaire (SF-MPQ): This questionnaire was used to establish the type of the dysmenorrhea pain in the subjects. The questionnaire consists of 15 items in 2 sub-scales that consist of the sensory (11 items) and affective pain (4 items) sub-scales. Each item is evaluated with a Likert-type scale between 0 and 3 (0: none, 3: severe), and the sum of these results established the total pain score. Furthermore, the evaluative total pain intensity index was measured using a 6-point Likert-type scale. In this scale '0' represents no detectable pain, whereas '5' represents unbearable pain. The Turkish version of the questionnaire was tested for its validity and reliability in 2007 and found to be reliable and valid.

The Depression Anxiety and Stress Scale (DASS): This scale was developed by Lovibond and Lovibond in 1995 to identify the emotional states of depression, anxiety and stress. The validity and reliability studies of its Turkish form were performed by Akın and Çetin in 2007. The scale includes 42 questions in which the given answers are evaluated quantitively between 0 (not suitable for me) and 3 (fully suitable for me). Depression, anxiety and stress are rated as normal, mild, moderate, advanced and extreme. This scale was included in the study to determine the effects of the heat treatment on depression, anxiety or stress.

Menstrual Attitude Questionnaire (MAQ): The reliability and the validity of the scale used to establish the attitudes and the behaviors of the subjects during menstruation were tested by Kulakaç et al. (2008). The scale includes 31 items as follows; menstruation as a debilitating event (7 items), menstruation as a bothersome event (5 items), menstruation as a natural event (5 items), anticipation and prediction of the onset of menstruation (8 items) and denial of the effects of menstruation (6 items). Each item is evaluated between 1 and 5 (1: I strongly disagree, 5: I strongly agree) using a 5-point Likert-type scoring.

ELIGIBILITY:
Inclusion Criteria:

* the ages of 18-30,
* being nulliparous,
* having a VAS score of 2 and higher,
* not having a systemic or chronic disease
* not using hormonal contraceptives.

Exclusion Criteria:

* using forms of analgesic and alternative treatments during the study
* experiencing menstrual irregularities

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
severity of dysmenorrhea assessed by Visual Analogue Scale | Change from Baseline severity of dysmenorrhea at 4 months
  Dysmenorrhea level, Visual Analog Scale The scale features a 10-cm long vertical line, with 0 at the bottom end and 10 at the top end

SECONDARY OUTCOMES:
Rate of Depression, Anxiety and Stress at Menstrual Cycle | İmmediately after the intervention at 4 Menstrual Cycle
  Depression Anxiety and Stress: The scale includes 42 questions in which the given answers are evaluated quantitively between 0 (not suitable for me) and 3 (fully suitable for me). Depression, anxiety and stress are rated as normal, mild, moderate, advanced and extreme. Higher scores mean a more severe depression, anxiety and stress
Rate of Menstrual Attitudes at Menstrual Cycle | İmmediately after the intervention at 4 Menstrual Cycle
  Menstrual Attitudes: The scale includes 31 items as follows; menstruation as a debilitating event (7 items), menstruation as a bothersome event (5 items), menstruation as a natural event (5 items), anticipation and prediction of the onset of menstruation (8 items) and denial of the effects of menstruation (6 items). Each item is evaluated between 1 and 5 (1: I strongly disagree, 5: I strongly agree) using a 5-point Likert-type scoring. higher scores mean a better Menstrual Attitudes

CONTACTS AND LOCATIONS:
Locations (1):
- Hülya TÜRKMEN, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No